CLINICAL TRIAL: NCT02403609
Title: An Online Study of the Reliability of the Brain Performance Test (BPT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lumos Labs, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: LL003
Record Dates: First submitted 2015-03-26; First posted 2015-03-31 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Healthy Volunteers
Keywords: cognitive assessment; Brain Performance Test; Lumosity; test-retest reliability; computerized assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BPT, Computerized Assessment (Experimental): Participants will first take the Brain Performance Test (BPT) on two consecutive days
  Interventions: Other: BPT, Computerized Assessment

INTERVENTIONS:
Other: BPT, Computerized Assessment

SUMMARY:
The purpose of this study is to evaluate test-retest reliability of each subtest (correlation coefficients for Time 1 and 2) in the Brain Performance Test (BPT, Lumos Labs, Inc.).

DETAILED DESCRIPTION:
This is an open-label, randomized online study in which participants will be invited to take versions of the Brain Performance Test (BPT) on two consecutive days.

In parallel, all current Lumosity subscribers are invited to take the BPT at the beginning of their premium Lumosity experience and again every 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Electronically signed informed consent
* English-speaker
* Current Lumosity free user (test-retest portion) OR current Lumosity subscriber (longitudinal portion)

Exclusion Criteria:

* Visual or physical impairment that impedes computer use or completion
* Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1357 (Actual)
Dates: Start 2015-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Correlation coefficients (Pearson's r) | 2 days
  Correlation coefficients (Pearson's r) of scaled scores of BPT subtests at Time 1 compared to Time 2

SECONDARY OUTCOMES:
Intercorrelation coefficients (Pearson's r) | 1 day
  Intercorrelation coefficients (Pearson's r) of scaled scores of BPT subtests at Time 1
Principle component analysis | 1 day
  Principle component analysis of scaled scores of BPT subtests at Time 1
Longitudinal BPT Grand Index and Subtest scaled scores | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Morrison, PhD, Principal Investigator — Lumos Labs, Inc.
Locations (1):
- Lumos Labs, Inc., San Francisco, California, United States

REFERENCES:
- See also: Click here for more information about Lumosity's Human Cognition Project. — http://www.lumosity.com/hcp/